CLINICAL TRIAL: NCT06636149
Title: CIRCUIT: Maternal Maneuvers During Prolonged Labor, a Pilot Randomized Control Trial
Brief Title: Maternal Maneuvers During Prolonged Labor
Acronym: CIRCUIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Drew Hensel, Physician, Fellow - Maternal Fetal Medicine, Barnes-Jewish Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202408190
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Labor Stage, First; Prolonged Labor
Keywords: Circuit; Position changes; Labor; Prolonged labor; Labor dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circuit Intervention Arm (Experimental): The intervention cohort will undergo the circuit of position changes every 2 hours. The circuit will be repeated up to 3 times or until the second stage of labor is achieved, delivery occurs, or labor arrest diagnosis is made. Participants will be considered as adherent to intervention arm if they undergo one complete circuit of maneuvers. Nurses will keep patients on continuous fetal monitoring during the circuit of position changes. Any persistent non-reassuring fetal status in one position of the circuit will prompt progression to the next position in the circuit. The planned circuit of maneuvers will be: 10-minutes of side-lying release on one side 10-minutes of side-lying release on other side 10-minutes of open-knee chest 10-minutes of shaking apples 20-minutes of flying cowgirl on one side 20-minutes of flying cowgirl on opposite side as position 5 20-minutes of running man on same side as position 5 20-minutes of running man on opposite side as position 5
  Interventions: Other: Circuit of maternal position changes during labor
- Control Arm (No Intervention): Patients randomized to the control arm will have their labor courses managed per current best practice recommendations. This will include nurse or patient facilitated position changes per the discretion of the patient's clinical care team. Routine position changes allowed in this control group will include walking, sitting, squatting, thrones, supine, hands and knees, and lateral decubitus with or without peanut ball. No positions in the circuit intervention group will be permitted to be used in the control group. Any circuit positions used in the control group will be tracked and documented.

INTERVENTIONS:
Other: Circuit of maternal position changes during labor — The intervention cohort will undergo the circuit of position changes every 2 hours. The circuit will be repeated up to 3 times or until the second stage of labor is achieved, delivery occurs, or labor arrest diagnosis is made. Participants will be considered as adherent to intervention arm if they undergo one complete circuit of maneuvers. Nurses will keep patients on continuous fetal monitoring during the circuit of position changes. Any persistent non-reassuring fetal status in one position of the circuit will prompt progression to the next position in the circuit. The planned circuit of maneuvers will be:
  10-minutes of side-lying release on one side 10-minutes of side-lying release on other side 10-minutes of open-knee chest 10-minutes of shaking apples 20-minutes of flying cowgirl on one side 20-minutes of flying cowgirl on opposite side as position 5 20-minutes of running man on same side as position 5 20-minutes of running man on opposite side as position 5
  Arms: Circuit Intervention Arm

SUMMARY:
This pilot, randomized control trial will test whether or not a specific circuit of position changes improves maternal outcomes in cases of prolonged labor.

Patient who have prolonged labor will be approached for consent and randomization to one of two study groups: circuit intervention against routine standard of care position changes. 82 patients will be enrolled in the study. Exclusion criteria will include: any uterine infection prior to randomization, magnesium sulfate treatment, major fetal anomalies, BMI ≥50, non-reassuring fetal status prior to randomization, or any maternal diagnosis that precludes safety or feasibility of the circuit of maternal position changes.

The 3 aims of the study will include: the outcome that the circuit of position changes has on the duration of the first stage of labor, maternal and neonatal morbidity, and maternal satisfaction.

DETAILED DESCRIPTION:
To date, there is an absence of data on intrapartum maternal position changes' efficacy or whether a specific circuit of intrapartum maneuvers is effective. We hypothesize that a nurse-informed circuit of positional maneuvers in protracted labor will significantly decrease the first stage of labor. The objective of this randomized control trial will be to assess whether a specific circuit of maternal position changes in prolonged latent or active labor will decrease the first stage of labor length. The three aims of this study are as follows: determine the effect of a nurse-led circuit of maternal position changes versus routine care on first stage of labor duration in patients with protracted labor. Compare maternal and neonatal outcomes among those with protracted labor who undergo a nurse-led circuit of maternal position changes vs routine standard of care. Compare maternal satisfaction, sense of control over labor process, and acceptability of a circuit of maternal position changes for those who undergo a nurse-led circuit of maternal position changes vs routine standard of care.

Across the country, there is an emphasis to reduce cesarean delivery rates with a specific focus on reducing rates of primary cesarean deliveries in nulliparous, term, singleton, and vertex pregnancies. The most common indication for a primary cesarean delivery is labor arrest. As a possible solution, there has been an increased utilization of maternal position changes during labor. In some cases, these are specifically used in cases of a prolonged first stage of labor. While these specific position changes are likely not associated with maternal or fetal harm, they require significant buy in from nursing and labor and delivery staff. Not only is increased time at the bedside required to execute these maneuvers, but they also often require multiple members of the care team, especially in patients with epidurals or obesity. To date, no study, retrospective or prospective, has evaluated the efficacy of a specific set of maternal maneuvers during prolonged first stage of labor. If a specific circuit of maternal maneuvers is found to decrease the first stage of labor duration in cases of protracted labor, then this would represent a significant intervention that could be offered to improve labor outcomes in patients.

This study's aim is to evaluate if, in cases of a prolonged first stage of labor, a specific circuit of maternal position changes leads to shorter first stage of labor duration. The study will be a prospective, randomized, pilot trial that will be conducted at Barnes Jewish Hospital in St. Louis, Missouri. This trial design was selected to minimize confounding factors and study the effects of a circuit of maternal position changes as specifically as possible. This trial will represent the first of its type to prospectively study the benefits of maternal position changes in cases of protracted labor.

This study's inclusion and exclusion criteria are listed later in this submission. Patients will be approached, enrolled, and consented to participate upon their admission to Labor and Delivery or when they have a diagnosis of protracted labor. Randomization will occur once they meet study criteria for protracted labor. Randomization will be done via a computer-generated block randomization sequence in a 1:1 ratio of the RN-led circuit of maternal maneuvers versus routine care during the remaining portion of the patient's labor course. Blinding will not be possible for the nursing team or physician team caring for patient. Data collection reviewers will be blinded to the participant's randomization arm.

Patients will be either randomized to routine care or a maternal circuit of labor position changes. These arms are described in detail later in the submission.

The type of maneuvers and specific order were created based on data from a nationwide survey for labor and delivery nurses regarding their personal experience and use of maneuver circuits. Compliance with the circuit of position changes and deviations from the planned circuit will be tracked.

Labor and delivery nurses will receive educational materials on how to perform the circuit of maternal position changes. The educational materials will remain available on labor and delivery for reference. Nursing stakeholders will serve as resources and provide assistance if any of their colleagues have issues with maneuvers on their shift.

The rest of labor induction and labor management will continue per standard of care. Oxytocin titration will be per our unit protocol. If the maximum oxytocin dose is reached, then consideration for oxytocin pausing and resumption will be at the primary provider's discretion. Oxytocin management data will be collected by research staff.

During the participant's postpartum stay, they will be approached to complete a maternal satisfaction survey regarding their labor experience, sense of control over the labor process, and circuit of position changes acceptability for those who underwent the intervention. The survey will be a brief, easily administered, 7-point Likert scale survey.

Our primary outcome will be first stage of labor duration. Secondary outcomes are listed later in this submission. Maternal surveys regarding satisfaction, sense of control over labor process, and acceptability for the circuit of maternal position changes will also be a secondary outcome.

Data on antenatal, intrapartum, and postpartum courses will be extracted from the medical record by a blinded investigator. This blinded investigator will also review the electronic medical record for pre-specified neonatal outcomes after delivery. Research staff will also monitor compliance with the assigned intervention and cross-over. Outcomes will be assessed from delivery until discharge.

Upon admission to labor and delivery or when diagnosis of protracted labor is made per study protocol, patients will be approached by trained research staff members to be enrolled in the study. This will be done in a private labor and delivery room. Research staff members will function independently and separately from the medical team caring for the patient. The patient will be given a brief introduction to the study, and if they are interested in learning more, the consent form will be reviewed in its entirety. Any questions will be answered by research staff. If, once their questions have been answered, the patient desires to participate, they and the research team member will sign and date the informed consent form. A copy will be given to the patient per standard protocol.

The principal investigator (PI) will review all adverse events. A data and safety monitoring board (DSMB) will also be established. This board will include three individuals not involved in the study. The PI will report all serious, adverse events to the DSMB within 72 hours of determination of occurrence. Reportable severe, adverse outcomes include intrauterine fetal demise after randomization, neonatal demise prior to maternal hospital discharge, or maternal death after randomization. Reportable non-severe adverse outcomes include intrapartum maternal fall or trauma during circuit maneuvers. Aside from maternal falls during circuit maneuvers, which we do not anticipate, all these adverse outcomes are not-study specific. All can occur, albeit rarely, because of labor and delivery complications or prolonged labor courses. We do not anticipate that study participation would increase any of these complications, but their incidence will be monitored. Non-severe events will be reported to the DSMB and IRB on an annual basis. Given the small sample size, no interim analyses will be performed as the study will not be powered to detect differences.

For data analysis, intention-to-treat and per-protocol analyses will be performed. Chi-squared and Fisher's exact tests will be used to compare categorical variables as appropriate. Continuous variables will be assessed for their distribution pattern using the Kolmogorov-Smirnov test. Normally distributed variables will be compared using the student's t-test and non-normally distributed variables will be analyzed with the Mann-Whitney U test. A Kaplan-Meier survival curve will also be used to evaluate the primary outcome. These analyses will be supplemented by multivariable logistic regressions to adjust for confounders. Results with p-values &lt;0.05 will be considered statistically significant. Analyses will be performed using Stata (Stata Corporation, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* Singleton, vertex pregnancies
* 34 weeks' gestation or later
* Admitted to Labor and Delivery in spontaneous labor or for an induction of labor
* Prolonged labor course as defined by: cervical dilation less than 6 cm after 8 hours or more of ruptured membranes (spontaneous or artificial) and oxytocin infusion, or cervical dilation 6 cm or more and less than 1-cm cervical dilation change over 2 hours or more with ruptured membranes and oxytocin infusion

Exclusion Criteria:

* Intraamniotic infection prior to randomization
* Magnesium sulfate treatment
* Major fetal anomalies
* BMI ≥50
* Non-reassuring fetal status prior to randomization
* Any maternal diagnosis that precludes safety or feasibility of intrapartum circuit of maternal position changes

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
First stage of labor duration | From enrollment until delivery
  Time from first cervical exam in spontaneous labor or first induction agent administration for induction of labor until patient has achieved cervical dilation of 10cm.

SECONDARY OUTCOMES:
Mode of delivery | Enrollment to delivery
  Type of delivery patient undergoes: vaginal delivery, operative vaginal delivery, or cesarean delivery
Cesarean section indication | Enrollment to delivery
  Reason patient underwent cesarean delivery
Length of labor | Enrollment to delivery
  Time from initial cervical exam for any patient admitted with spontaneous labor or time from first induction agent administration for inductions of labor until delivery
Length of active labor | Time from 6cm of cervical dilation to 10cm of cervical dilation or delivery
  Time from cervical exam of 6cm or more until patient has cervical dilation of 10cm or delivery
Length of latent labor | Admission until active labor (cervix 6cm or greater) or delivery
  Time from initial cervical exam for any patient admitted with spontaneous labor or time from first induction agent administration for inductions of labor until cervical exam with dilation of 6cm or more, or undergoes delivery.
Length of second stage of labor | 10cm of cervical dilation to delivery
  Time from cervical dilation of 10cm until delivery
Time from randomization to delivery | Time from randomization to delivery
  Time from when patient randomized into study until delivery
Time from randomization to second stage of labor | Time from randomization until patient achieves 10cm cervical dilation
  Time from randomization until patient achieves 10cm cervical dilation
Composite maternal morbidity | Enrollment to postpartum discharge
  Includes: postpartum hemorrhage, maternal blood transfusion, severe perineal laceration (3rd and 4th degree), ICU admission, and maternal death
Composite Neonatal Morbidity | From delivery until neonatal discharge or 1 month of life (whichever comes first)
  Includes: neonatal death, respiratory distress defined as need for respiratory support within 72 hours after birth and consisting of one or more of the following: the use of continuous positive airway pressure (CPAP) or high-flow nasal cannula for at least 2 consecutive hours, supplemental oxygen with a fraction of inspired oxygen of at least 0.30 for at least 4 continuous hours, extracorporeal membrane oxygenation (ECMO), or mechanical ventilation, hypoxic-ischemic encephalopathy, intraventricular hemorrhage grade 3 or 4, necrotizing enterocolitis, 5 minute APGAR score <7, umbilical artery pH ≤7.1

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Medicine, Saint Loius, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carbonne B, Benachi A, Leveque ML, Cabrol D, Papiernik E. Maternal position during labor: effects on fetal oxygen saturation measured by pulse oximetry. Obstet Gynecol. 1996 Nov;88(5):797-800. doi: 10.1016/0029-7844(96)00298-0. PMID 8885916
- [Background] Gupta JK, Sood A, Hofmeyr GJ, Vogel JP. Position in the second stage of labour for women without epidural anaesthesia. Cochrane Database Syst Rev. 2017 May 25;5(5):CD002006. doi: 10.1002/14651858.CD002006.pub4. PMID 28539008
- [Background] Roberts JE, Mendez-Bauer C, Wodell DA. The effects of maternal position on uterine contractility and efficiency. Birth. 1983 Winter;10(4):243-9. doi: 10.1111/j.1523-536x.1983.tb01433.x. No abstract available. PMID 6556913
- [Background] Mendez-Bauer C, Arroyo J, Garcia Ramos C, Menendez A, Lavilla M, Izquierdo F, Villa Elizaga I, Zamarriego J. Effects of standing position on spontaneous uterine contractility and other aspects of labor. J Perinat Med. 1975;3(2):89-100. doi: 10.1515/jpme.1975.3.2.89. PMID 1185484
- [Background] Tussey CM, Botsios E, Gerkin RD, Kelly LA, Gamez J, Mensik J. Reducing Length of Labor and Cesarean Surgery Rate Using a Peanut Ball for Women Laboring With an Epidural. J Perinat Educ. 2015;24(1):16-24. doi: 10.1891/1058-1243.24.1.16. PMID 26937158
- [Background] Hickey L, Savage J. Effect of Peanut Ball and Position Changes in Women Laboring With an Epidural. Nurs Womens Health. 2019 Jun;23(3):245-252. doi: 10.1016/j.nwh.2019.04.004. Epub 2019 May 9. PMID 31077640
- [Background] Harvey S, Rach D, Stainton MC, Jarrell J, Brant R. Evaluation of satisfaction with midwifery care. Midwifery. 2002 Dec;18(4):260-7. doi: 10.1054/midw.2002.0317. PMID 12473441
- [Background] McCoy JA, Walheim L, McCabe MG, Levine LD. Efficacy of Propranolol to Reduce Cesarean Delivery in Prolonged Labor: A Randomized Controlled Trial. Obstet Gynecol. 2023 Jul 1;142(1):71-79. doi: 10.1097/AOG.0000000000005232. Epub 2023 Jun 7. PMID 37290102